CLINICAL TRIAL: NCT05537545
Title: A Randomized Controlled Trial on the Timing of Soft Tissue Grafting Following Immediate Implant Placement
Brief Title: Timing of Soft Tissue Grafting Following Immediate Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2022-0258
Record Dates: First submitted 2022-09-01; First posted 2022-09-13 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Bone Resorption
Keywords: dental implant, single tooth; immediate; connective tissue graft
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: As this RCT concerns a surgical intervention, patients and treating clinicians can not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate soft tissue grafting (Active Comparator): A connective tissue graft is immediately harvested and inserted in the buccal mucosa at the moment of implant placement
  Interventions: Procedure: Soft tissue grafting
- Delayed soft tissue grafting (Experimental): Three months after implant placement, a connective tissue graft is harvested and inserted in the buccal mucosa
  Interventions: Procedure: Soft tissue grafting

INTERVENTIONS:
Procedure: Soft tissue grafting — A pouch is made in the buccal mucosa using microsurgical instruments. Thereupon, a free gingival graft is harvested from the palatal mucosa in the premolar area and de-epithelialized to arrive at a CTG of about 1 mm thickness. Height and length are tailored to the dimensions of the site. Then, the CTG is brought into the pouch and fixed with two single sutures (Seralon 6/0, Serag Wiessner, Naila, Germany) onto the buccal mucosa.

SUMMARY:
Patients undergoing single immediate implant placement (IIP) in the premaxilla will be invited to participate in this randomized controlled trial (RCT). Prior to surgery, a small- field low-dose cone beam computed tomography (CBCT) is taken to verify the integrity of the facial bone wall and an adequate amount of apical and palatal bone availability for implant anchorage.

In all of the patients, a connective tissue graft (CTG) will be harvested and inserted into the buccal mucosa to increase soft tissue thickness around the immediately installed implant. However, included patients will be randomly allocated to either receive the CTG immediately after implant installation (Immediate soft tissue grafting, ISG = control group) or 3 months after implant installation (Delayed soft tissue grafting, DSG = test group).

Forty sealed envelopes are prepared for that purpose, of which 20 are internally labeled as "DSG" and 20 as "ISG". Following IIP, a sealed envelope will be opened to reveal the treatment concept In both groups, a cutting implant is installed in an optimal 3D position. Socket grafting is performed with deproteinized bovine bone mineral to limit buccal bone resorption and to optimize soft tissue stability.

In the ISG group, a pouch is made in the buccal mucosa using microsurgical instruments. Thereupon, a free gingival graft is harvested from the palatal mucosa in the premolar area and de-epithelialized to arrive at a CTG of about 1 mm thickness. Height and length are tailored to the dimensions of the site. Then, the CTG is brought into the pouch and fixed with two single sutures onto the buccal mucosa. Finally, a healing abutment is installed, which is replaced by a provisional implant crown 2 days later.

In the DSG group, implant placement, socket grafting and installation of a provisional implant crown occur as described above. In contrast, a buccal pouch is performed 3 months after implant installation. Graft harvesting, adaptation and fixation are performed as described above.

A small-field low-dose CBCT is taken at the 1-year and 5-year follow-up in order to measure buccal bone resorption as compared to the baseline dimensions in designated software.

DETAILED DESCRIPTION:
Patients with a single failing tooth in the anterior maxilla will be included after a clinical examination and evaluation of a small-field low-dose CBCT. An intra-oral scan will be taken in order to make a surgical guide. A cutting implant with variable thread design (BLX, Straumann) will be installed using the surgical guide in order to sufficient primary implant stability.

Thereafter, the gap between the implant surface and buccal bone wall is filled with deproteinized bovine bone mineral (Bio-Oss, Gheistlich Pharma).

At this point, a closed envelope is opened and the patient gets assigned to either ISG or DSG group.

In the immediate soft tissue grafting group, a de-epithelialized free gingival graft was inserted in a buccal pouch to augment the buccal soft tissues. The graft was fixed with single sutures (Seralon 6/0, Serag Wiessner, Naila, Germany).

In the delayed soft tissue grafting group, the same procedure was performed 3 months after implant placement.

In both groups, patients received an immediate, screw-retained temporary crown. Restorations were installed within the first 48h after implant placement.

Sutures were removed 1 week after soft tissue grafting.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years old
* Good oral hygiene defined as full-mouth plaque score ≤ 25% (O'Leary et al. 1972)
* Presence of an incisor, cuspid or premolar in the maxilla that needs to be extracted for any reason with at least one neighboring tooth present
* At least 3 mm bone available at the apical or palatal aspect of the alveolus as assessed on CBCT to ensure primary implant stability
* Intact buccal bone wall at the time of extraction
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Systemic diseases
* Smoking
* Suppuration
* > 1 mm gingival asymmetry between the failing and contralateral tooth
* Untreated periodontal disease; untreated caries lesions

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Buccal bone resorption (mm) | 1-, 5-year
  Changes in buccal bone dimension as measured on superimposed CBCT slides

SECONDARY OUTCOMES:
Changes in buccal soft tissue profile (mm) | 1-, 5-year
  Changes in buccal soft tissue profile as measured on superimposed digital surface models. An intra-oral scan is taken prior to implant surgery and at 1- and 5- year follow up. On the obtained digital models, an area of interest (AOI) at the buccal aspect was drawn for each site. The AOI extends from 0.5 mm below the soft tissue margin to 4 mm more apical. In mesio-distal dimension, the AOI reaches from the mesial to the distal line angle. The AOI may vary between sites because of individual anatomic differences but must be kept constant in each site across time points. A volumetric change (mm3) was calculated by designated software within the AOI and divided by the AOI surface (mm2). This results in the mean change in buccal soft tissue profile (mm).
Changes in midfacial soft tissue level (mm) | 1-, 5-year
  Changes in buccal mucosal margin position as measured on superimposed digital surface models
Pink Esthetic Score | 1-year
  Pink Esthetic score as defined by Fürhauser et al., 2005. Within this scale, 7 variables are evaluated ( mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture) using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value, the maximum achievable PES was 14. A 0 relates to the least esthetic result, while a 14 relates to a perfect outcome for all parameters.
Mucosal Scarring Index | 1-year
  Mucosal Scarring Index as defined by Wessels et al., 2019. Within this scale, 5 parameters are assessed (width, height/contour, color, suture marks, and overall appearance) using a 0-1-2 scoring system. The MSI score may range from 0 (no scar) to 10 (most extreme scar).
Marginal bone level changes (mm) | 1-,5-year
  Changes in the distance from the implant-abutment interface to the first bone-to-implant contact (so-called marginal bone level) at the mesial and distal aspect of each implant as measured on 2D intra-oral radiographs
Probing depth (mm) | 1-,5-year
  Measured with a periodontal probe at four locations (mesio-buccal, buccal, disto-buccal and oral) around the implant at 1- and 5-year follow-up. Measurements are rounded up to the nearest 0.5 mm. A mean value is calculated per implant.
Plaque (%) | 1-,5-year
  Presence of plaque at four locations (mesio-buccal, buccal, disto-buccal and oral) around the implant. Each location is scored 0 or 1
Bleeding on probing (%) | 1-,5-year
  Presence of bleeding on probing at four locations (mesio-buccal, buccal, disto-buccal and oral) around the implant. Each location is scored 0 or 1

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Zuiderveld EG, van Nimwegen WG, Meijer HJA, Jung RE, Muhlemann S, Vissink A, Raghoebar GM. Effect of connective tissue grafting on buccal bone changes based on cone beam computed tomography scans in the esthetic zone of single immediate implants: A 1-year randomized controlled trial. J Periodontol. 2021 Apr;92(4):553-561. doi: 10.1002/JPER.20-0217. Epub 2020 Sep 11. PMID 32918332
- [Background] Seyssens L, Eghbali A, Christiaens V, De Bruyckere T, Doornewaard R, Cosyn J. A one-year prospective study on alveolar ridge preservation using collagen-enriched deproteinized bovine bone mineral and saddle connective tissue graft: A cone beam computed tomography analysis. Clin Implant Dent Relat Res. 2019 Oct;21(5):853-861. doi: 10.1111/cid.12843. Epub 2019 Aug 28. PMID 31456345
- [Background] Wessels R, De Roose S, De Bruyckere T, Eghbali A, Jacquet W, De Rouck T, Cosyn J. The Mucosal Scarring Index: reliability of a new composite index for assessing scarring following oral surgery. Clin Oral Investig. 2019 Mar;23(3):1209-1215. doi: 10.1007/s00784-018-2535-6. Epub 2018 Jul 3. PMID 29971512
- [Derived] Struys T, Christiaens V, De Bruyckere T, Pitman J, Van Hove PJ, Cosyn J. A Randomized Controlled Trial on the Timing of Soft Tissue Augmentation in Immediate Implant Placement: Soft Tissue Changes and Esthetic Outcome. Clin Implant Dent Relat Res. 2025 Feb;27(1):e70013. doi: 10.1111/cid.70013. PMID 39980395
- [Derived] Cosyn J, Struys T, Van Hove PJ, De Buyser S, De Bruyckere T. A Randomized Controlled Trial on the Timing of Soft-Tissue Augmentation in Immediate Implant Placement: Hard-Tissue Changes and Clinical Outcome. J Clin Periodontol. 2024 Nov;51(11):1534-1544. doi: 10.1111/jcpe.14060. Epub 2024 Sep 1. PMID 39218777